CLINICAL TRIAL: NCT03864705
Title: Compliance of Diabetic Patients Treated With Metformin
Acronym: CODAMET
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Institute for Clinical and Experimental Medicine (Other Government)
Responsible Party: Principal Investigator, Martin Haluzik, Clinical Scientist, Institute for Clinical and Experimental Medicine
Other Study IDs: 001
Record Dates: First submitted 2019-03-03; First posted 2019-03-06 (Actual); Last update posted 2020-09-11 (Actual); Status verified 2020-09

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Measurement of plasma metformin levels — Subjects on chronic metformin therapy will have their plasma metformin levels measured during a regular check-up with glycated hemoglobin assessment.

SUMMARY:
Metformin is the 1st line treatment in all subjects with type 2 diabetes without a contraindication to its use. The compliance with the use of metformin is not optimal mainly owing to relatively frequent gastrointestinal side effects. However, hard data about the real compliance are currently not available.

In this trial we aim at assessing the compliance with metformin intake using a combination of serum metformin measurement and a specific questionnaire. We will further evaluate the impact of different pharmacological forms of metformin (standard vs. XR - extended release) on its compliance and try to identify common characteristics associated with reduced compliance.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus on metformin therapy for at least 3 months

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with type 2 diabetes mellitus on metformin therapy for at least 3 months.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Plasma metformin levels | At the time of measurement

CONTACTS AND LOCATIONS:
Overall Officials: Martin Haluzik, Prof. DSc., Principal Investigator — Institute for Clinical and Experimental Medicine
Locations (1):
- Institute for Clinical and Experimental Medicine, Prague, Czechia

IPD SHARING:
Plan to Share IPD: No